CLINICAL TRIAL: NCT02450864
Title: The Biological Effect of Extracorporeal Shockwave Technology (ESWT) and the Role of Proinflammatory Cytokines and Cannabinoid Receptor in Shoulder Stiffness
Brief Title: The Biological Effect of ESWT and the Role of Proinflammatory Cytokines and Cannabinoid Receptor in Shoulder Stiffness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: IRB 101-1810A3
Record Dates: First submitted 2015-04-13; First posted 2015-05-21 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Stiffness of Shoulder, Not Elsewhere Classified
Keywords: Stiffness of Shoulder, Not Elsewhere Classified

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patient with ESWT (Experimental): Preoperatively, the ROM of the shoulder is measure with the patient in a sitting position. A goniometer is used to measure the angle to which the patient could maximally passively forward flex or abduct the shoulder. External rotation and internal rotation of the shoulders are determined with the patient's arm in a resting position. The investigators assessed shoulder ROM using the SROMD. Normal shoulder ROM without scapular stabilization is considered to be 180° of forward flexion, 180° of abduction, 90° of external rotation, and 90° of internal rotation with the arm at the side. By summation of the measured deficit of ROM, the SROMD is obtained. Patients are defined as having shoulder stiffness if SROMD >270degrees.
  Interventions: Other: ESWT
- patient without ESWT (Sham Comparator): Preoperatively, the ROM of the shoulder is measure with the patient in a sitting position. A goniometer is used to measure the angle to which the patient could maximally passively forward flex or abduct the shoulder. External rotation and internal rotation of the shoulders are determined with the patient's arm in a resting position. The investigators assessed shoulder ROM using the SROMD. Normal shoulder ROM without scapular stabilization is considered to be 180° of forward flexion, 180° of abduction, 90° of external rotation, and 90° of internal rotation with the arm at the side. By summation of the measured deficit of ROM, the SROMD is obtained. Patients are defined as having shoulder stiffness if SROMD >270degrees.
  Interventions: Other: ESWT

INTERVENTIONS:
Other: ESWT — Preoperatively, the ROM of the shoulder is measure with the patient in a sitting position. A goniometer is used to measure the angle to which the patient could maximally passively forward flex or abduct the shoulder. External rotation and internal rotation of the shoulders are determined with the patient's arm in a resting position. The investigators assessed shoulder ROM using the SROMD. Normal shoulder ROM without scapular stabilization is considered to be 180° of forward flexion, 180° of abduction, 90° of external rotation, and 90° of internal rotation with the arm at the side. By summation of the measured deficit of ROM, the SROMD is obtained. Patients are defined as having shoulder stiffness if SROMD >270degrees.

SUMMARY:
Investigators recent data showed anti-inflammatory effect of Effect of Extracorporeal Shockwave Technology (ESWT). Little studies focused on the effect and pathomechanism of ESWT on shoulder stiffness.

DETAILED DESCRIPTION:
1. First year:Investigators intend to further delineate the inflammatory mechanism, such as IL-1β, CB1, HSP in the incidence of shoulder stiffness.
2. Second year: Investigators intend to conduct a prospective randomized double-blind study for the clinical effect of ESWT on patients with shoulder stiffness.
3. Third year: Investigators wish to test the biologic effect of ESWT on patients with shoulder stiffness and to elucidate the molecular mechanism for this effect through a randomized comparative study.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 80 years
* receiving surgery for open acromioplasty

Exclusion Criteria:

* shoulder disorders caused by traumatic fracture
* previous surgery
* osteoarthritis
* malignant disorders
* hepatic disorders
* renal disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-01-01; Primary Completion 2019-07-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
the range of motion (ROM) of the shoulder as a measure | 1weeks
  Preoperatively, the ROM of the shoulder is measure with the patient in a sitting position. A goniometer is used to measure the angle to which the patient could maximally passively forward flex or abduct the shoulder. External rotation and internal rotation of the shoulders are determined with the patient's arm in a resting position. The investigators assessed shoulder ROM using the SROMD. Normal shoulder ROM without scapular stabilization is considered to be 180° of forward flexion, 180° of abduction, 90° of external rotation, and 90° of internal rotation with the arm at the side. By summation of the measured deficit of ROM, the SROMD is obtained. Patients are defined as having shoulder stiffness if SROMD >270degrees.

CONTACTS AND LOCATIONS:
Overall Officials: Jih-Yang Jih-Yang, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung City, Taiwan